CLINICAL TRIAL: NCT06023160
Title: Predicting Functional Outcome and Response to Therapy of Anti-NMDAR Encephalitis at Diagnosis: The NEOSII Score
Brief Title: Predicting Functional Outcome and Response to Therapy of Anti-NMDAR Encephalitis at Diagnosis
Acronym: NEOSII
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Maarten J. Titulaer. MD, PhD, Associate professor, Dr., Erasmus Medical Center
Other Study IDs: NEOSII
Record Dates: First submitted 2023-08-19; First posted 2023-09-05 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Anti-NMDA (N-Methyl D-Aspartate) Receptor Encephalitis
Keywords: Prognosis; Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Dutch National anti-NMDAR Encephalitis Cohort: Dutch National anti-NMDAR Encephalitis Cohort
- German anti-NMDAR Encephalitis Cohort (GENERATE): German anti-NMDAR Encephalitis Cohort (GENERATE)
- Spanish anti-NMDAR Encephalitis Cohort: Spanish anti-NMDAR Encephalitis Cohort
- French anti-NMDAR Encephalitis Cohort: French anti-NMDAR Encephalitis Cohort
- Japanese anti-NMDAR Encephalitis Cohort: Japanese anti-NMDAR Encephalitis Cohort

SUMMARY:
The goal of this international cohort study is to develop a prediction model for long-term outcome and response to first-line immunotherapy of anti-NMDAR Encephalitis, already at the moment of diagnosis.

DETAILED DESCRIPTION:
Anti-NMDARE is a severe, but treatable neurological condition, with considerable and variable long-term disability. The previously developed anti-NMDAR Encephalitis One-Year Functional Status (NEOS) score predicts outcome a month into treatment. To predict outcome and response to immunotherapy at the time of diagnosis would be a serious improvement. This would timely identify patients in need for aggressive treatment and avoid harmful side-effects in those with good outcome. International data from five anti-NMDAR encephalitis cohorts will be combined to attain these goals.

The investigators strive to have less than 10% missing data on all variables and will impute data were needed. The datasets will then be split - with equal distributions of cohorts and good/poor outcome - to develop (70%) and validate (30%) the NEOS2 model. The primary outcome is functioning one year after diagnosis. A secondary analysis is targeted to predict the effect of first-line therapy. Potentially relevant predictive variables are identified with a univariable analysis on the original data, confirmed with backwards selection on the imputed datasets. After checking for multicollinearity and linearity of the variables, identified variables are added to a mixed effects logistic regression model on the original and imputed datasets, to identify the final set of predictive variables. To make the models opportune for daily medical practice, the investigators will assign points to (categories of) the included variables, based on the coefficients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with anti-NMDAR encephalitis (according to the Graus criteria)

Exclusion Criteria:

* Preceding Herpes Simplex encephalitis
* Premorbid dependency (modified Rankin Scale > 2)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective data of five (inter)national anti-NMDAR encephalitis cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 714 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Functional status one year after diagnosis, on the modified Rankin Scale. | One year after diagnosis
  The score on the modified Rankin Scale will be applied as the original ordinal scale as well as dichotomized, where scores 0-2 represent "independent functioning" (without or with symptoms) and scores 3-6 increasing levels of depencency

SECONDARY OUTCOMES:
Response to first-line immunotherapy | Two weeks after administration of first-line immunotherapy
  One point improvement (one point lower than at diagnosis) on the modified Rankin Scale (ranging from 0 - no symptoms - to 6 - deceased - as the most severe category) within two weeks from therapy commencement.
Return to school or work | Throughout follow-up time after diagnosis (different per patient, depending on date of diagnosis). Average 3 years (min 0 - max 22 years)
  Time-to-event analysis on the ability to return to school or work during follow-up, including timing of resumption of work after diagnosis.
Relapse rate | Throughout follow-up time after diagnosis (different per patient, depending on date of diagnosis). Average 3 years (min 0 - max 22 years)
  Time-to-event analysis on relapses during total available follow-up time, including time of relapse after diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten J. Titulaer, Assoc. Porf., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands